CLINICAL TRIAL: NCT03450200
Title: Effectiveness of Exercises in Patient With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Mi Mi Thet Mon Win, Graduate Student, Okayama University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D16-07; Ethics/DMR/2017/048 (Other: Department of Medical Research, Myanmar)
Record Dates: First submitted 2018-02-19; First posted 2018-03-01 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy, Exercises
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises Group (Experimental): three times daily exercises of hands and fingers exercises and foot exercises which last for 10 minutes in eight weeks, and health education about diabetic foot care
  Interventions: Other: exercises for diabetic peripheral neuropathy; Other: Health education for diabetic foot care
- Control Group (Other): health education about diabetic foot care
  Interventions: Other: Health education for diabetic foot care

INTERVENTIONS:
Other: exercises for diabetic peripheral neuropathy — Hands, fingers, and foot exercises for diabetic peripheral neuropathy to improve activities of daily living, and decreases the signs and symptoms of DPN
  Arms: Exercises Group
Other: Health education for diabetic foot care — Health education for daily diabetic foot care to prevent diabetic foot ulcer was provided.

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is the common complication seen in the diabetic patients. Moreover, it will lead to another complication as disabilities and difficulties in activities of daily living (ADL). Most of the intervention for diabetes and diabetic neuropathic patients are mostly focusing on the prevention of foot ulcer. Diabetic foot care can prevent only for diabetes-related foot ulcer and foot amputation. It cannot be reduced DPN and cannot be improved the activities of daily living of the patient with DPN. Moreover, there is the restriction of weight-bearing exercise on the recommendation of exercises for the patients with DPN. Therefore, exercise program which may be suitable for all the patients with DPN was introduced in this study to improve ADL and decrease the neuropathic symptoms in the diabetic patients.

Compliance with exercise or intervention is not only critical to get adherence but also for the long-term use of its. Easy to do exercise in the short duration which can able to do on their own in their home promote their compliance and adherence to the exercises. In this study, the effectiveness of exercises in the patients with diabetic peripheral neuropathy was examined to fulfill the requirement of exercises which is simple and can be done in a short time. The objective of the study is to examine the effectiveness of exercise in the patients with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* The patients receiving diabetic care at the out-patient-department of designated hospitals, able to contact via the telephone, presence of signs and symptoms of DPN, agreed to involve in the study (informed consent), and aged over 25 years

Exclusion Criteria:

* The persons who are suffering from DPN other than diabetes, severe illness of diabetic patients, diabetes with other comorbidities, amputation of hands and feet from any reasons, mental illness and alcoholism

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Change in Activities of daily living (ADLs) after intervention, at follow-up | eight weeks after intervention, eight weeks follow-up
  ADLs were measured by using Patient Neurotoxicity Questionnaire (PNQ).
Change in signs of DPN after intervention, at follow-up | eight weeks after intervention, eight weeks follow-up
  DPN was assessed by using monofilament (SMW), Touch-TestTM Sensory Evaluator 5 Pieces Hand Kit of North Coast Medical Inc.
Change in signs of DPN after intervention, at follow-up | eight weeks after intervention, eight weeks follow-up
  DPN was assessed by tuning fork vibration test.

SECONDARY OUTCOMES:
Change in strength of hand grip | eight weeks after intervention, eight weeks follow-up
  Hand grip was measured in kilograms by using TTM original Dynamometer 100 kg.
Change in strength of pinch force | eight weeks after intervention, eight weeks follow-up
  Key (lateral pinch) was measured by the gold standard B&L Engineering® Pinch Gauge 0-30 lb. in 1.0 lb.
Change in walking speed | eight weeks after intervention, eight weeks follow-up
  Timed Up and Go (TUG) test was to measure the duration for walking in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Mi Thet Mon Win, PhD student, Principal Investigator — Graduate School of Health Sciences, Okayama University
Locations (1):
- Okayama University, Okayama, Japan